## **Informed Consent Form**

Version No. 0.2\_en, 21.05.2024

Title of the Study: ColoReg: A Register for Findings and Videos of Endoscopies in Gastroenterology

Name of the patient in block letters: .....

| • | I have been informed by about the nature, significance, and scope of |
|---|---|
| | the study as well as the requirements that arise for me from it. I have also read the text of the patient information and this consent form. |
| • | I had sufficient time to ask questions and make a decision. Any questions that arose were answered by the study doctor. |
| | I know that I can end my voluntary participation at any time without any disadvantages aris- |
| | ing for me. |
| | I consent to participate in the study. |
| • | • |
| • | I consent to the collection of personal data about me, particularly video material and find- |
| | ings from the examination, as described in the information sheet, and to the recording and |
| | temporary processing of this data in paper form and on electronic media at the treating cen- |
| | ter, in this case at the University Hospital Würzburg. |
| • | The collected data may be shared and published in anonymized form as described in the |
| | patient information. |
| • | I also consent to the study initiator, who is bound to confidentiality, reviewing the collected |
| | study data in individual cases, as far as necessary to verify anonymization. |
| • | I have been informed that my data will be published in anonymized form for teaching and |
| | research purposes. I have been informed that I cannot participate in this study without of |
| | senting to the publication of my data in anonymized form. |
| • | I have been informed that I can revoke my consent at any time. In the event of revocation, |
| | no further data will be collected. After inclusion in the study, your data will be available in |
| | pseudonymized form for at least 3 months, and up to 12 months if follow-up is planned. If |
| | such data is available at the time of revocation, it will be deleted immediately. I had addi- |
| | tional questions: |

- I had the opportunity to ask questions and received answers.
- I had sufficient time to decide to participate in the project.
- I have received a copy of the patient information and consent form.
- I consent to participate in the research project and the associated processing of the mentioned data.

Studie: ColoReg Einwilligungserklärung, Versions Nr.: 0.2, 21.05.2024

• I have received a copy of the information sheet and consent form. One copy remains at the study center.

| Signature of the participant | |
|------------------------------------------------------|-------------|
| (Name and first name in block letters) | |
| (Date) (Signature) | |
| Declaration and signature of the informing doct | or: |
| I conducted the information session and obtained the | ne consent. |
| (Name and first name in block letters) | |
| (Date) (Signature) | |